CLINICAL TRIAL: NCT05831748
Title: The Effects of Clinical Pilates Training on Balance and Walking in Lower Limb Prosthesis Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Albina Alikaj, Principal Investigator, Medipol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-2675
Record Dates: First submitted 2023-04-03; First posted 2023-04-26 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Prosthesis User
Keywords: pilates; gait analyses; balance; prosthesis; amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 15 Transfemoral and Transtibial amputees will be included in this group. Patients will be treated with classic physiotherapy exercises for 12 weeks. Patients will practice exercises 3 times a week, one time in clinics with a physiotherapist and 2 times as home exercise.
  Interventions: Other: Classic Exercise
- Active Comparator group (Active Comparator): 15 Transfemoral and Transtibial amputees will be included in this group. Patients will be treated with Clinical pilates exercises for 12 weeks. Patients will practice exercises 3 times a week, one time in clinics with a physiotherapist and 2 times as home exercise.
  Interventions: Other: Clinical Pilates

INTERVENTIONS:
Other: Classic Exercise — Classic exercise group consists of straight leg raising, back extensor strengthening, and abdominal strengthening exercises.
  Arms: Experimental Group
Other: Clinical Pilates — In the Clinical pilates group, pilates exercises will be given. Clinical pilates exercises improve back extensors, trunk flexors, and pelvis stabilization. These exercises will be applied along with breathing exercises.
  Arms: Active Comparator group

SUMMARY:
Studies have shown that Pilates exercises are one of the exercises that can improve breathing capacity, coordination, balance, flexibility, and muscular endurance. Pilates exercises improve walking and balance, reduce back pain and prevent further pain or injury. These are all common problems for people who have undergone lower extremity amputation. The aim of our study is to improve the pelvis-trunk coordination, gait symmetry, and balance on individuals who have undergone amputation and also to increase body awareness.

DETAILED DESCRIPTION:
The patients will be randomly assigned to two groups. Clinical Pilates (CP) and Classic Physiotherapy (CF). Two groups will be Transfemoral and Transtibial amputees, one CP, and the other CF. Groups will be treated for a period of 12 weeks. The assessment will be made before the treatment and after 12 weeks. Patients will practise exercises 3 times a week, one time in clinics with a physiotherapist and 2 times as home exercise.

In the clinical Pilates group, exercises that improve back extensor, trunk flexor, and pelvis stabilization will be applied along with breathing exercises. The classic group consists of straight leg raising, back extensors strengthening, abdominal strengthening exercises.

Gait spatiotemporal parameters, balance, fall risk and mobility, functional capacity, core muscle endurance, and strength, the pain will be evaluated. Quality of life, body image, and also prosthesis satisfaction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Be a Volunteer,
* Being at least 6 months after amputation,
* Having no problems related to prostheses,
* Using a hydraulic, pneumatic, or microprocessor knee joint type,
* According to the functional classification of amputees, individuals at the K3-K4 level,
* Individuals with unilateral transtibial, unilateral transfemoral amputation

Exclusion Criteria:

* Users using assistive devices,
* Those with bilateral amputation,
* Those having contractures,
* Those with acute low back pain,
* Spine and lower extremity involvement due to systemic inflammation (rheumatoid arthritis, spondyloarthropathy, etc.),
* Systemic neurological disease (Multiple sclerosis, Alzheimer's, etc.),
* Patients with other diseases that prevent mobilization (vertigo, cerebellar ataxia, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Gait analyses | 10 Minutes
  Basic gait parameters include walking speed, step length and cadence will be evaluated.

SECONDARY OUTCOMES:
The tandem walk test (TWT) | 1 minute
  The tandem walk test (TWT) is a physical performance test used to assess balance and coordination. During the TWT, the individual is asked to walk a straight line, placing the heel of one foot directly in front of the toes of the other foot. This creates a "tandem" or heel-to-toe gait. The individual is instructed to take as many steps as possible along the line without stepping off or losing balance. The TWT is typically performed over a distance of 3-5 meters, and the time it takes the individual to complete the test is recorded.
Berg Balance Scale | 20 minutes
  The Berg Balance Scale (BBS) is a widely used clinical assessment tool that is used to measure an individual's ability to maintain balance during different functional tasks. The BBS consists of 14 different tasks that assess different aspects of balance, including sitting unsupported, standing unsupported, transferring from sitting to standing, standing with eyes closed, standing with feet together, turning 360 degrees, reaching forward, retrieving objects from the floor, and stepping up and down on a stool.
  Each task is scored on a 5-point scale, with a maximum score of 56 points. The scores for each task are summed to obtain a total score, which provides a measure of the individual's overall balance performance. Higher scores indicate better balance performance, while lower scores indicate greater difficulty maintaining balance.
Six Minute Walk Test | 6 minutes
  The 6-minute walk test (6MWT) is a simple and widely used clinical tool to assess the exercise capacity and functional status of a person. It involves measuring the distance a person can walk on a flat surface in 6 minutes at their own comfortable pace.
  The general steps involved in performing a 6MWT:
  The person is given instructions on how to perform the test, which includes walking as far as they can within 6 minutes without running.
  The person is allowed to rest for a short period of time (usually 10-15 minutes) before the test begins.
  The person is asked to walk back and forth along a marked 30-meter course or a long hallway.
  The person's oxygen saturation level, heart rate, and blood pressure are monitored before and after the test.
  The total distance covered by the person in 6 minutes is measured. The test will be performed in a controlled environment, such as a clinic, and is supervised by a specialised physiotherapist.
Core muscle endurance test | 1-3 minutes
  The core muscle endurance test is a measure of the endurance of the muscles of core, which includes your abdominal muscles, back muscles, and pelvic muscles. The test is typically used to evaluate core strength and muscular endurance. To perform the core muscle endurance test, a timer and a mat is needed. These steps should be followed:
  Lie down on your back on the mat with your arms at your sides and your knees bent.
  Lift your feet off the ground so that your knees are at a 90-degree angle. Raise your head and shoulders off the mat, keeping your chin tucked and your neck relaxed.
  Hold this position for as long as you can, keeping your knees at a 90-degree angle and your feet off the ground.
  Stop the timer when you can no longer maintain the position or when your form begins to suffer.
  The test measures the time you can hold this position, with longer times indicating greater core muscle endurance. A good score for the test varies depending on age, sex, and fitness level.
SF-36 (Short Form 36) | 5-10 minutes
  SF-36 (Short Form 36) is a questionnaire used to measure health-related quality of life. Shorter version of the SF-12 questionnaire and contains 36 questions that assess eight health concepts, including physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Albina Alikaj, PhD(c), Principal Investigator — Medipol University; Esra Atılgan, Assoc.Prof., Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Varrecchia T, Serrao M, Rinaldi M, Ranavolo A, Conforto S, De Marchis C, Simonetti A, Poni I, Castellano S, Silvetti A, Tatarelli A, Fiori L, Conte C, Draicchio F. Common and specific gait patterns in people with varying anatomical levels of lower limb amputation and different prosthetic components. Hum Mov Sci. 2019 Aug;66:9-21. doi: 10.1016/j.humov.2019.03.008. Epub 2019 Mar 16. PMID 30889496
- [Result] den Otter AR, Geurts AC, Mulder T, Duysens J. Speed related changes in muscle activity from normal to very slow walking speeds. Gait Posture. 2004 Jun;19(3):270-8. doi: 10.1016/S0966-6362(03)00071-7. PMID 15125916
- [Result] Ulger O, Yildirim Sahan T, Celik SE. A systematic literature review of physiotherapy and rehabilitation approaches to lower-limb amputation. Physiother Theory Pract. 2018 Nov;34(11):821-834. doi: 10.1080/09593985.2018.1425938. Epub 2018 Jan 19. PMID 29351504
- [Result] Asano M, Rushton P, Miller WC, Deathe BA. Predictors of quality of life among individuals who have a lower limb amputation. Prosthet Orthot Int. 2008 Jun;32(2):231-43. doi: 10.1080/03093640802024955. PMID 18569891
- [Result] Esquenazi A. Gait analysis in lower-limb amputation and prosthetic rehabilitation. Phys Med Rehabil Clin N Am. 2014 Feb;25(1):153-67. doi: 10.1016/j.pmr.2013.09.006. PMID 24287245